CLINICAL TRIAL: NCT01110369
Title: A Protein Supplementation and Exercise Strategy to Promote Muscle Protein Anabolism in Frail Elderly People
Acronym: ProMuscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lisette de Groot, Professor, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1002-2
Record Dates: First submitted 2010-02-12; First posted 2010-04-26 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia
Keywords: sarcopenia; frail elderly; protein drink; resistance exercise; Skeletal muscle mass; muscle mass in elderly
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance exercise training and protein drink (Experimental)
  Interventions: Dietary Supplement: Protein drink; Other: Resistance exercise training
- Resistance exercise training and placebo drink (Placebo Comparator)
  Interventions: Other: Resistance exercise training; Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Protein drink — Protein drink twice a day during 6 months.
  Arms: Resistance exercise training and protein drink
Other: Resistance exercise training — Resistance exercise training twice per week during 6 months.
Dietary Supplement: Placebo drink — Placebo drink twice a day during 6 months.
  Arms: Resistance exercise training and placebo drink

SUMMARY:
The present study is designed to investigate whether timed protein supplementation will increase skeletal muscle mass in the frail elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly individuals
* Able to understand and perform the study procedures

Exclusion Criteria:

* Type I or type II diabetes (fasted blood glucose level ≥7,0 mmol)
* No recent history (within 2 years) of participating in any regular resistance exercise training program (general questionnaire)
* Use of anti-coagulation medication (except of Acetyl Salicyl acid)
* Presence of coronary heart disease (ECG)
* Renal insufficiency (eGFR <60 mL/min/1.73 m2)
* Allergic or sensitive for milk proteins

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle mass | Baseline, 3 months and 6 months

SECONDARY OUTCOMES:
Physical performance | Baseline, 3 months and 6 months
Blood will be collected to assess parameters related to the outcome measures | Baseline, 3 months and 6 months
Dietary intake | Baseline, 3 months and 6 months
Physical activity | Baseline, 3 months and 6 months
Cognitive performance | Baseline and 6 months
Blood pressure | Baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Professor, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Dorhout BG, de Groot LCPGM, van Dongen EJI, Doets EL, Haveman-Nies A. Effects and contextual factors of a diet and resistance exercise intervention vary across settings: an overview of three successive ProMuscle interventions. BMC Geriatr. 2022 Mar 9;22(1):189. doi: 10.1186/s12877-021-02733-6. PMID 35264105
- [Derived] van de Rest O, van der Zwaluw NL, Tieland M, Adam JJ, Hiddink GJ, van Loon LJ, de Groot LC. Effect of resistance-type exercise training with or without protein supplementation on cognitive functioning in frail and pre-frail elderly: secondary analysis of a randomized, double-blind, placebo-controlled trial. Mech Ageing Dev. 2014 Mar-Apr;136-137:85-93. doi: 10.1016/j.mad.2013.12.005. Epub 2013 Dec 27. PMID 24374288
- [Derived] Tieland M, Dirks ML, van der Zwaluw N, Verdijk LB, van de Rest O, de Groot LC, van Loon LJ. Protein supplementation increases muscle mass gain during prolonged resistance-type exercise training in frail elderly people: a randomized, double-blind, placebo-controlled trial. J Am Med Dir Assoc. 2012 Oct;13(8):713-9. doi: 10.1016/j.jamda.2012.05.020. Epub 2012 Jul 6. PMID 22770932